CLINICAL TRIAL: NCT04445805
Title: The INSPIRE Trial: Improving Negative Stressful Perseverations in Insomnia to Revitalize Expectant Moms
Brief Title: Improving Negative Stressful Perseverations in Insomnia to Revitalize Expectant Moms
Acronym: INSPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, David Kalmbach, Bioscientific Staff Researcher, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INSPIRE
Record Dates: First submitted 2020-06-19; First posted 2020-06-24 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Insomnia
Keywords: Insomnia; Telemedecine; pregnancy; perinatal; Cognitive Arousal; depression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBTI Treatment Group (Active Comparator): Telemedicine Cognitive Behavioral Therapy for Insomnia (CBTI)
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBTI)
- Perinatal-enhanced behavioral therapy for insomnia (Experimental): Telemedicine Mindfulness Based Therapy for Insomnia (MBTI)
  Interventions: Behavioral: Perinatal-enhanced Behavioral Therapy for Insomnia
- Attention Control Treatment Group (Placebo Comparator): Minimal intervention control
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBTI) — Consists of 6 prenatal 60-min sessions and 6 monthly postnatal sessions on sleep education, sleep restriction, stimulus control, cognitive therapy, and relaxation. Treatment will be delivered via telemedicine.
  Arms: CBTI Treatment Group
Behavioral: Perinatal-enhanced Behavioral Therapy for Insomnia — Consists of 6 prenatal 60-min sessions and 6 monthly postnatal sessions on sleep education, sleep restriction, stimulus control, and metacognitive exercises. Treatment will be delivered via telemedicine.
  Arms: Perinatal-enhanced behavioral therapy for insomnia
Behavioral: Attention Control — Will include education on sleep, circadian rhythms, and good sleep hygiene in addition to self-monitoring with sleep diaries.
  Arms: Attention Control Treatment Group

SUMMARY:
The purpose of this research is to evaluate telemedicine treatments for sleep in pregnant women. As pregnant women are vulnerable to sleep problems, the investigators aim to explore whether these types of treatment will improve sleep and mood-related health risks in pregnancy and postpartum. The investigators will test the efficacy of cognitive behavioral therapy for insomnia (CBTI) and mindfulness-based therapy for insomnia (MBTI) for perinatal insomnia relative to sleep education and hygiene, which is a minimal intervention control.

DETAILED DESCRIPTION:
The purpose of this randomized controlled trial is to determine the efficacy of cognitive behavioral therapy for insomnia (CBTI) and mindfulness-based therapy for insomnia (MBTI) for perinatal insomnia relative to sleep education and hygiene, which is a minimal intervention control. The long-term goal is to maximize the effectiveness of insomnia treatment for perinatal women by adapting safe and efficacious treatments to meet the evolving needs of women through pregnancy and postpartum. Over half of pregnant women develop insomnia, which is associated with high rates of depression during pregnancy and postpartum. By successfully treating insomnia during pregnancy and improving cognitive-emotion regulation, mental health of pregnant and postpartum women may be substantially improved. In a prior clinical trial, Dr. Kalmbach (PI) showed that digital CBTI (i.e., fully automated online program) improved sleep during pregnancy, and offered some protection against sleep problems after childbirth. Women in this prior trial were highly satisfied with CBTI and the ability to participate in treatment remotely. However, the investigators identified important shortcomings of CBTI in this population. Namely, standard CBTI was ineffective at reducing cognitive arousal and depression. Preliminary data suggest that MBTI may effectively reduce cognitive arousal in insomnia patients, which has immense potential to enhance sleep and mental health outcomes in perinatal insomnia. Thus, the investigators will conduct a randomized controlled trial to determine the efficacy of MBTI and CBTI for perinatal insomnia relative to a minimal intervention control.

The current study is a 3-arm RCT comparing CBTI and MBTI to sleep education and hygiene minimal intervention control for the treatment of perinatal insomnia. 120 women with insomnia symptoms will be treated beginning in pregnancy and into early postpartum. CBTI and MBTI will address changes in sleep symptoms and challenges that emerge after childbirth. The investigators will collect outcome data on insomnia symptoms and related health outcomes (e.g., cognitive arousal, depression) after prenatal treatment and monthly across the first postpartum year. The investigators will determine the efficacy of the investigator's CBTI and MBTI protocols for perinatal insomnia relative to minimal intervention control. The investigators will then compare the effects of CBTI and MBTI on short- and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* (1) Gestational age at time of study enrollment must be less than or equal to 28 weeks
* (2) Insomnia Severity Index score > 10
* (3) age 18 - 40 years
* (4) reliable and adequately fast internet connection at home, which is required to engage in telemedicine treatment (online video) and online study outcome assessments.

Exclusion Criteria:

* High risk pregnancy (e.g., pre-eclampsia, multiple pregnancy, age>40)
* Bipolar disorder (contraindicated for CBTI)
* Seizures (contraindicated for CBTI)
* Active suicidal intent
* Shift work
* Patients who cannot reasonably engage in study activities including treatment or completing online surveys will be excluded regardless of reason. This may include inability to comprehend the English language, inability to hear therapist over video sessions, inability to understand and meaningfully answer study outcomes measures, or other barriers to participation.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness of mindfulness based therapy for insomnia for changes in insomnia symptoms - Insomnia Severity Index (ISI) | Will be assessed pretreatment, immediately posttreatment, and monthly across the 1st postnatal year
  The Insomnia Severity Index (ISI) is a commonly used self-report measure of insomnia symptoms that has been validated for use in community samples and clinical trials. The ISI scores range from 0-28, with a higher score indicating a greater severity of insomnia. ISI scores < 8 after treatment indicate remission.

SECONDARY OUTCOMES:
Effectiveness of mindfulness based therapy for insomnia for changes in depression symptoms- Edinburgh Postnatal Depression Scale (EPDS) | Will be assessed pretreatment, immediately posttreatment, and monthly across the 1st postnatal year
  The Edinburgh Postnatal Depression (EPDS) is the most widely used depression measure in both pregnant and postnatal women. It is validated for use in community samples and clinical trials. The EPDS scores range from 0-30, with a higher score indicating a greater severity of depression.
Effectiveness of mindfulness based therapy for insomnia for changes in cognitive arousal - Presleep Arousal Scale-Cognitive Factor | Will be assessed pretreatment, immediately posttreatment, and monthly across the 1st postnatal year
  The Presleep Arousal Scale- Cognitive Factor is a commonly used self-report measure of nocturnal cognitive arousal that has been validated for use in community samples and clinical trials. The scores range from 8-40, with a higher score indicating a greater severity of nocturnal cognitive arousal.

CONTACTS AND LOCATIONS:
Overall Officials: David Kalmbach, PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Medical Center, Novi, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided